CLINICAL TRIAL: NCT02899416
Title: Better Life by Nutrition During Adulthood : Identification of Factors Present in Adolescence Cardiovascular Risk in Young Adults
Brief Title: Better Life by Nutrition During Adulthood
Acronym: BELINDA
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2015_24; 2016-A00386-45 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-08-24; First posted 2016-09-14 (Estimated); Last update posted 2025-12-23 (Actual); Status verified 2022-09

CONDITIONS: Cardiovascular Risk Factor
Keywords: cardiovascular risk; young adulthood

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA used for telemore length
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
BELINDA is a follow'up of subjects included 10 years ago in HELENA study which was a cross-sectional study carried out from 2006 to 2007 in more than 3500 adolescents aged from 12.5 to 17.5 years old through 10 Europeans towns from 9 countries.

BELINDA main objective is to assess CV risk using PDAY score (Pathobiological Determinants of Atherosclerosis in Youth) during young adulthood (20 to 31 years) and analyze lifestyle risk factors from adolescence (12 to 18 years). This analyze may define new CV risk factors and risk population cluster.

DETAILED DESCRIPTION:
BELINDA subjects from Lille, Ghent , Zaragoza and Roma will be re-tested using a part of HELENA test battery and some new evaluation criteria.

ELIGIBILITY:
Inclusion Criteria:

* Women of men participating to HELENA study 2006-2007
* Aged from 20 to 35 years.
* Signed informed consent

Exclusion Criteria:

* Pregnant or lactating women

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: BELINDA is a follow'up of subjects included 10 years ago in HELENA study which was a cross-sectional study carried out from 2006 to 2007 in more than 3500 adolescents aged from 12.5 to 17.5 years old through 10 Europeans towns from 9 countries.
  BELINDA will retest subjects from Lille and Ghent
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
PDAY score (Pathobiological Determinants of Atherosclerosis in Youth) | one day
  PDAY score is a composite score which will be calculated using adult data including Gender, HDL non cholesterol, HDL cholesterol. Glucose level, Blood pressure, Tobacco consumption and BMI.

SECONDARY OUTCOMES:
Diet Quality Index Score | 2 days
  data collected using HELENA-DIAT, an electronic dietary recall, data in DQI score unit.
  DQI score is ranking from 0 to 9 unit and is based on three basic principles for a healthy diet: quality; diversity; balance. Furthermore, the daily diet was divided into nine recommended food groups, namely (1) water, (2) bread and cereals, (3) grains and potatoes, (4) vegetables, (5) fruit, (6) milk products (7), cheese, (8) meat, fish, eggs and substitutes, and (9) fats and oils.
Ratio total energy intake | 2 days
  data collected using HELENA-DIAT, an electronic dietary recall, data in kcal/d, data for recommended total energy intake will be collected using national reference chart.
ratio of dietary n-6/n-3 polyunsaturated fatty acids (PUFA) | 2 days
  data collected using HELENA-DIAT, an electronic dietary recall, data in ratio calculated using a food composition data base. PUFA is expressed in mg/day daily intake.
consumption in dietary salt intake | 2 days
  data collected using HELENA-DIAT, an electronic dietary recall, data in mg/day daily intake calculated using a food composition data base.
Physical activity | 7 days
  data collected using a GT3X accelerometer data in daily counts/min
Endurance | 1 day
  data collected using Dr Leger Shuttle run test, data in VO2max ml/kg/min
Ratio waist-to-hip | 1 day
  data collected using anthropometric measurements, data in ratio. Data are expressed in centimeter
Fat mass | 1 day
  data collected using anthropometric measurements, data in % of fat mass, expressed in kg
Education level | 1 day
  data collected using a Socio-economic questionnaire, data in Education level 8 digits

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Gottrand, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHRU,Hôpital Jeanne de Flandres, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Morcel J, Beghin L, Michels N, De Ruyter T, Drumez E, Cailliau E, Polito A, Le Donne C, Barnaba L, Azzini E, De Henauw S, Miguel Berges ML, Cacau LT, Moreno LA, Gottrand F. Nutritional and physical fitness parameters in adolescence impact cardiovascular health in adulthood. Clin Nutr. 2024 Aug;43(8):1857-1864. doi: 10.1016/j.clnu.2024.06.022. Epub 2024 Jun 26. PMID 38959665